CLINICAL TRIAL: NCT02842307
Title: Impact of Acupuncturist Expertise on Clinical Effectiveness for Chemotherapy Induced Nausea and Vomiting in Cancer Patients: a Randomized Controlled Trial
Brief Title: Acupuncture for Chemical Therapy Induced Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yutong Fei, Associate research fellow, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBM@BUCM-2; 30901929 (Other Grant/Funding Number: National Natural Science)
Record Dates: First submitted 2016-07-16; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Acupuncture; Expertise-based randomized controlled trial; Nausea; Vomiting; Cancer
MeSH Terms: conditions — Vomiting; Nausea; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A(senior acupuncturists) (Active Comparator): Manual acupuncture implemented by senior acupuncturists (clinical experience >15 years)
  Interventions: Procedure: Manual acupuncture implemented by senior acupuncturists
- B(junior acupuncturists) (Active Comparator): Manual acupuncture implemented by junior acupuncturists (clinical experience <5 years)
  Interventions: Procedure: Manual acupuncture implemented by junior acupuncturists
- C(P6 points) (Active Comparator): Manual acupuncture on P6 points by junior acupuncturists (clinical experience <5 years)
  Interventions: Procedure: Manual acupuncture on P6 point
- D(no acupuncture) (No Intervention): No acupuncture treatment

INTERVENTIONS:
Procedure: Manual acupuncture implemented by senior acupuncturists — Manual acupuncture once per day. No limitation on points, manipulations and time per session. Senior acupuncturists have to have more than 15 years of acupuncture clinical practice experience.
  Other Names: Traditional manual acupuncture; Traditional acupuncture
  Arms: A(senior acupuncturists)
Procedure: Manual acupuncture implemented by junior acupuncturists — Manual acupuncture once per day. No limitation on points, manipulations and time per session. Junior acupuncturists have to have less than 5 years of acupuncture clinical practice experience.
  Other Names: Traditional manual acupuncture; Traditional acupuncture
  Arms: B(junior acupuncturists)
Procedure: Manual acupuncture on P6 point — Manual acupuncture implemented by junior acupuncturists once per day. P6 point, bilaterally, should achieve deqi sensation by even manipulations. Junior acupuncturists have to have less than 5 years of acupuncture clinical practice experience.
  Other Names: Traditional manual acupuncture; Traditional acupuncture
  Arms: C(P6 points)

SUMMARY:
This is an expertise-based randomized controlled trial. The hypothesis of this study is that the differences in expertise of acupuncturist may impact clinical effect. In this study, patients will be randomized to 4 group, receiving the treatment from senior acupuncturist, junior acupuncturist, junior acupuncturist by only acupuncture Neiguan(P6), or not receive the acupuncture. All patients receive the basic cisplatin chemotherapy. The duration of treatment is from the first day receiving cisplatin until two days after cisplatin on each group. NCI and Rhode scale will be used to measure the control of nausea and vomiting.

DETAILED DESCRIPTION:
This is an expertise-based randomized controlled trial. The hypothesis of this study is that the differences in expertise of acupuncturist may impact clinical effect. In this study, 102 patients will be randomly divided into 4 groups which separately receiving the treatment from senior acupuncturist(clinical experience> 15 years, considered in this trial as highly expertised), junior acupuncturist(clinical experience< 5 years, considered in this trial as lower expertised), junior acupuncturist only acupuncture Neiguan(P6), or not receiving the acupuncture. All participants receive the cisplatin-based chemotherapy and 5-HT3 as antiemetic treatment will be included. Acupuncture treatments are given once daily, the duration of treatment is from the first day receiving cisplatin until two days after cisplatin. NCI and Rhode scale will be used to measure the control of nausea and vomiting. only outcome assessors are blinded. Generalized estimating equations will be used to compare the effects among groups.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cancer
* Must receive cancer chemotherapy containing cisplatin
* Use 5-TH receptor antagonists as an antiemetic drug in the chemotherapy duration

Exclusion Criteria:

* Concurrent neoplasms or illness that induces nausea independent of chemotherapy
* Received acupuncture treatments for other conditions less than 4 weeks before chemotherapy treatment
* Severe infection
* Severe heart, liver, kidney and brain diseases
* Cardiac pacemaker
* Radiotherapy or hormone therapy during chemotherapy treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
NCI nausea and vomiting rating scale | From the first day receiving cisplatin until two days after cisplatin in each group
Rhodes Scale | From the first day receiving cisplatin until two days after cisplatin in each group

SECONDARY OUTCOMES:
Global assessment on effectiveness by patients (a single direct question with five levels of alternatives) | The second day after cisplatin
Patients' confidence towards acupuncture treatment (a single direct question with five levels of alternatives) | The first day receiving cisplatin and the second day after cisplatin
Consumption of additional antiemetic | From the first day receiving cisplatin until two days after cisplatin

OTHER OUTCOMES:
Acupuncture related adverse events | From the first day receiving cisplatin until two days after cisplatin
Adverse events | From the first day receiving cisplatin until two days after cisplatin

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Dongzhimen Hospital, Beijing University of Chinese medicine, Beijing, Beijing Municipality
  - Guanganmen Hospital,China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing